CLINICAL TRIAL: NCT06065852
Title: National Registry of Rare Kidney Diseases (RaDaR)
Brief Title: National Registry of Rare Kidney Diseases
Acronym: RaDaR
Status: Recruiting | Type: Observational
Sponsor: UK Kidney Association (Other)
Responsible Party: Sponsor
Other Study IDs: RaDaR
Record Dates: First submitted 2023-09-19; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Adenine Phosphoribosyltransferase Deficiency; AH Amyloidosis; AHL Amyloidosis; AL Amyloidosis; Alport Syndrome; Atypical Hemolytic Uremic Syndrome; Autoimmune Distal Renal Tubular Acidosis; Autosomal Recessive Proximal Renal Tubular Acidosis; Autosomal Recessive Distal Renal Tubular Acidosis; Autosomal Dominant Polycystic Kidney Disease; Autosomal Recessive Polycystic Kidney Disease; Bartter Syndrome; BK Nephropathy; C3 Glomerulopathy With Monoclonal Gammopathy; C3 Glomerulopathy; Calciphylaxis; Crystalglobulinaemia; Crystal-storing Histiocytosis; Cystinosis; Cystinuria; Dense Deposit Disease; Dent Disease; Denys-Drash Syndrome; Dominant Hypophosphataemia With Nephrolithiasis and/or Osteoporosis; Drug Induced Fanconi Syndrome; Drug-Induced Hypomagnesemia; Drug-Induced Nephrogenic Diabetes Insipidus; Epilepsy, Ataxia, Sensorineural Deafness and Tubulopathy; Fabry Disease; Familial Hypomagnesemia With Hypercalciuria and Nephrocalcinosis; Familial Primary Hypomagnesemia With Hypocalcuria; Familial Primary Hypomagnesaemia With Normocalciuria; Familial Renal Glucosuria; Fanconi Renotubular Syndrome 1; Fanconi Renotubular Syndrome 2; Fanconi Renotubular Syndrome 3; Fibrillary Glomerulonephritis; Fibromuscular Dysplasia; Focal Segmental Glomerulosclerosis; Generalised Pseudohypoaldosteronism Type 1; Gitelman Syndrome; Heavy-Metal-Induced Fanconi Syndrome; Hepatocyte Nuclear Factor 1-Beta-Associated Monogenic Diabetes; Hereditary Renal Hypouricemia; Hereditary Hypophosphatemic Rickets With Hypercalciuria; Hyperuricaemic Nephropathy; IgA Nephropathy; Immunotactoid Glomerulonephritis With Organised Microtubular Mononoclonal Immunoglobulin Deposits; Inherited Renal Cancer Syndromes; Intracapillary Monoclonal IgM Without Cryoglobulin; Intraglomerular/Capillary Lymphoma/Leukaemia; Isolated Autosomal Dominant Hypomagnesaemia Glaudemans Type; Liddle Syndrome; Light Chain Cast Nephropathy; Light Chain Proximal Tubulopathy Without Crystals; Light Chain Proximal Tubulopathy With Crystals; Lowe Syndrome; Membranous Nephropathy; Membranoproliferative Glomerulonephritis; Medullary Cystic Kidney Disease; Minimal Change Nephropathy; Mitochondrial Disease Of The Kidney; Monoclonal Immunoglobulin Deposition Disease; Nail Patella Syndrome; Nephrogenic Diabetes Insipidus; Nephrogenic Syndrome of Inappropriate Antidiuresis; Nephronophthisis; Primary Hypomagnesemia With Secondary Hypocalcemia; Primary Hyperoxaluria; Proliferative Glomerulonephritis With Monoclonal IgG Deposits; Proximal Tubulopathy Without Crystals; Pseudohypoaldosteronism Type 1, 2A-2E; Pure Red Cell Aplasia; Retroperitoneal Fibrosis; Sickle Cell Nephropathy; Shiga Toxin Associated Haemolytic Uraemic Syndrome; Steroid Resistant Nephrotic Syndrome; Steroid-Sensitive Nephrotic Syndrome; Thin Basement Membrane Nephropathy; Thrombotic Microangiopathy With Monoclonal Gammopathy; Type 1 Cryoglobulinaemic Glomerulonephritis; Tuberous Sclerosis; Unclassified Monoclonal Gammopathy Of Renal Significance; Vasculitis
MeSH Terms: conditions — Adenine phosphoribosyltransferase deficiency; Immunoglobulin Light-chain Amyloidosis; Nephritis, Hereditary; Atypical Hemolytic Uremic Syndrome; Renal tubular acidosis, distal, autosomal recessive; Polycystic Kidney, Autosomal Dominant; Polycystic Kidney, Autosomal Recessive; Bartter Syndrome; Calciphylaxis; Cystinosis; Cystinuria; Glomerulonephritis, Membranoproliferative; Dent Disease; Denys-Drash Syndrome; SeSAME syndrome; Fabry Disease; Hypomagnesemia primary; Hypomagnesemia 1, Intestinal; Glycosuria, Renal; Fibromuscular Dysplasia; Glomerulosclerosis, Focal Segmental; Gitelman Syndrome; Renal cysts and diabetes syndrome; Hypophosphatemic Rickets with Hypercalciuria, Hereditary; Glomerulonephritis, IGA; Liddle Syndrome; Oculocerebrorenal Syndrome; Glomerulonephritis, Membranous; Nephronophthisis, familial juvenile; Nephrosis, Lipoid; Nail-Patella Syndrome; Diabetes Insipidus, Nephrogenic; Nephrogenic Syndrome of Inappropriate Antidiuresis; Hyperoxaluria, Primary; Pseudohypoaldosteronism; Red-Cell Aplasia, Pure; Retroperitoneal Fibrosis; Nephrotic Syndrome; Hematuria, Benign Familial; Tuberous Sclerosis; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — RaDaR participants agree for their past, present and future clinical data to be used for ongoing and future research into kidney disease and related conditions. Some of this research involves the collection, processing and storage of biospecimens, including DNA. Individuals consent for this on an individual study basis.

GROUPS / COHORTS (31):
- Alport Syndrome Rare Disease Group: The evidence base in Alport Syndrome is small, but there is a very important education gap which it is the group's priority.
  Our first priorities are to assemble and make available clear information for clinicians caring for patients, as well as for patients themselves including making it clear for Commissioners 'Who should be tested' establish contact details for advice on specific issues make it clear how to approach the group for clinical advice and how to enrol patients in the group.
  In time this may lead to specialised regional clinics, made possible by recruiting more interested clinicians as the project develops.
- APRT Deficiency Rare Disease Group: Aims:
  1. To collect clinical data on patients with APRT Deficiency in a Registry. This will allow us to:
     study the causes, natural history and outcome of the condition develop patient cohorts for future studies
  2. To collect biological samples for future studies in a Biobank. This will allow us to:
     identify factors influencing the course of APRT Deficiency determine the role of various genes
  3. To develop new methods to measure urinary purine excretion. This will improve tools that allow us to:
     study the effectiveness of pharmacological and dietary interventions identify factors influencing the course of the condition
  4. To work with patient organisations, health care professionals and researchers:
  to enhance the education and training aspect of this project to develop strategies to increase the awareness and early detection of APRT Deficiency and improve patient outcomes.
- ARPKD & NPHP Rare Disease Group: Aims:
  The Autosomal Recessive Polycystic Kidney Disease (ARPKD)/Nephronophthisis (NPHP) Rare Disease Group (RDG) aims to:
  Develop and advocate best practice guidelines for the treatment of ARPKD and NPHP Provide up-to-date, best practice patient information and group support Support research into basic science, genetic, translational, psychosocial and clinical aspects of ARPKD and NPHP Foster collaborations with European and international groups and partner
- Atypical Haemolytic Uraemic Syndrome Rare Disease Group: Aims:
  To establish and maintain a registry of all individuals affected by aHUS in the UK To provide information to clinicians on the investigation and management of aHUS To provide information to affected individuals and their families on aHUS To facilitate collaborative research into all aspects of aHUS
- Autosomal Dominant Polycystic Kidney Disease Rare Disease Group: Aims:
  To develop the ADPKD RaDaR registry To develop best practice guidelines in regards to the treatment of ADPKD To provide better patient information and support To develop international collaborations to enable the above aims To support research, in collaboration with international groups, into basic science, disease progression models and clinical trials
- Autosomal Dominant Tubulointerstitial Kidney Disease Rare Disease Group: The group was established as part of the RaDaR initiative, in light of the increasing numbers of families being identified with this syndrome and following the pioneering work undertaken by Dr Anne Simmonds and others in the Purine Laboratory at Guy's Hospital, London.
- BK Nephropathy Rare Disease Group: The BK Nephropathy (BKN) Rare Disease Group aims to:
  collate contemporary information from UK kidney transplant recipients with BK Nephropathy use this information to develop current and relevant information for patients disseminate this information to the renal and transplant communities establish a national consensus to identify recipients at high risk of developing BK Nephropathy develop a recommendation for the optimal screening frequency for the presence of BK viraemia by PCR of peripheral blood produce guidance on the modification of immunosuppressive regimens and use of additional agents to treat BK Nephropathy develop a strategy for patient recruitment to observational and interventional clinical trials
- Calciphylaxis rare Disease Group: The Calciphylaxis Rare Disease Group aims to:
  Develop a comprehensive clinical database of Calciphylaxis patients via the RaDaR Rare Disease Registry Collaborate with international registries, particularly the German registry Form an expert panel of interested clinicians to review future clinical trials and research programmes Develop diagnostic and treatment algorithms
- CKD due to Genetic Factors in people of African ancestry Rare Disease Group: People of African or Afro-Caribbean ancestry are five times more likely to have kidney disease. They also develop kidney failure when they are about ten years younger than white people. The connection between ethnicity and kidney disease is complex. There have been some new scientific discoveries which may help us to begin to understand the cause of this problem and develop treatments, but much more work is needed.
  This group will allow us to find lots of people with African or Afro-Caribbean ancestry with CKD living in the UK that can take part in research.
- Cystinosis Rare Disease Group: Aims:
  To improve the care for all patients with cystinosis in the UK To collaborate with the National Designation Centres for Cystinosis To work together with Cystinosis Foundation UK and other patient groups To register every willing patient with cystinosis onto RaDaR To promote research for the benefit of patients with cystinosis, and their families To promote educational resources for patients with cystinosis, and their families
- Cystinuria Rare Disease Group: To improve our understanding of kidney stone formation in Cystinuria, develop best practice in the care of patients with this condition and to develop new ways to prevent and treat Cystinuria.
- Dent Disease & Lowe Syndrome Rare Disease Group: The group aims to advance our knowledge of Dent Disease and Lowe Syndrome by:
  establishing a registry of patients developing clinical guidelines regarding diagnosis and treatment providing a platform for clinical and molecular research into these disorders empowering affected patients and their families by facilitating contacts between patient/families and by the development of educational material
- Fabry Disease Rare Disease Group: The main objectives of the Fabry Disease Rare Disease Group are to:
  Provide reliable information for patients and relatives regarding the condition Provide referral information for clinicians, including details about where to send samples Improve referral pathways between the relevant specialties in each geographical area e.g. cardiology and nephrology Design and implement studies to determine the burden of undiagnosed disease and make testing for Fabry more accessible nationwide Organise patient information days to promote face-to-face contact between clinicians and patients/families
- Fibromuscular Dysplasia Rare Disease Group: The main objectives of the Fibromuscular Dysplasia Rare Disease Group are to:
  Raise awareness and provide advice about the best strategy for the diagnosis and management of this still underdiagnosed disease.
  Study the presentation of the disease and baseline patient demographics. Study the prevalence of different subtypes of Fibromuscular Dysplasia, the incidence and determinants of disease progression/extension and complications Develop a Register of long term impact of intervention, as part of RaDaR
- Haemolytic Uraemic Syndrome Rare Disease Group: 1. To identify key issues and challenges facing the field of Haemolytic Uraemic Syndrome, specifically in the development of an informatics framework within the UK
  2. To stimulate and encourage industry partnerships.
  3. To identify the needs and priorities for basic, clinical, translational and social research
  4. To identify suitable funding opportunities and help support appropriate strategies for successful applications.
- Hepatic Nuclear Factor 1B Mutation Rare Disease Group: The HNF1B rare disease group (RDG) covers all diseases associated with mutations and deletions in this gene. These include renal developmental disorders, most commonly renal cysts. The most common problem outside the kidneys is diabetes. When diabetes and renal cysts occur together this is known as the renal cysts and diabetes (RCAD) syndrome. Other clinical features may include hyperuricaemia and gout, hypomagnesaemia, abnormal liver function tests, pancreatic exocrine deficiency and genital tract malformations.
  We aim to increase clincians' awareness of these presentations, improve recognition and streamline diagnosis, particularly at a genetic level. To do this we are studying genetic information on patients with well-defined clinical features. We hold open meetings to inform and support patients and their families.
- Hyperoxaluria Rare Disease Group: The Hyperoxaluria Rare Disease Group aims to:
  The Hyperoxaluria Rare Disease Group aims to:
  Provide up to date support for patients and their families. Increase the knowledge and understanding of Primary Hyperoxaluria and Oxalosis to improve its clinical management.
  Provide clinical information on dialysis and transplantation. Increase the knowledge of clinical presentation and outcome of Primary Hyperoxaluria.
  Foster national and international partnerships to promote scientific innovation and research in Primary Hyperoxaluria and facilitate applications for funding for research collaboration.
  Create a forum for UK clinical studies on Primary Hyperoxaluria, including trials with orphan drugs.
  Foster genotype studies on Primary Hyperoxaluria. Co-operate in order to obtain funding for research activities through industrial or public partners in order to facilitate the dissemination of the results deriving from scientific research.'
- IgA Nephropathy Rare Disease Group: The IgA Nephropathy (IgAN) Rare Disease Group aims to:
  collate avaliable information on IgAN and develop new information for both patients and carers implement a communications strategy for the wider renal community about all aspects of the RDG's work programme develop a strategy for patient recruitment to clinical trials in IgAN
- Inherited Renal Cancer Syndromes Rare Disease Group: The development of evidence based clinical care pathways in inherited RCC has been identified as a priority owing to the lack of fully commissioned screening programmes nationally. Several published expert led disease management guidelines are being evaluated. Therefore the familial RCC RDG will set as a priority the development and validation of evidence based care pathways that reflect both national and international opinion and can be adopted by NHS commissioning groups.
  The familial RDG will work closely with other RDGs, the Renal Registry and the Renal Association to produce advice for commissioners that relate to specific aspects of these diseases as well as more general advice that relates to rare diseases, CKD and renal replacement therapy.
- Lupus Nephritis Rare Disease Group
- Membranous Nephropathy Rare Disease Group: Aims:
  1. To develop evidence based clinical care pathways. Current treatment for Membranous Nephropathy (MN) is based on knowledge and drugs available in the 1990's.
  2. To empower and inform patients and families.
  3. To audit clinical outcomes:
     Establish a registry of biopsy proven prevalent cases and new incident cases of both primary and secondary MN starting from Jan 2013. In total we seek to capture data on 2000 patients during the next 5 years with a minimum of one complete data return per patient per year.
  4. To promote and develop research.
- Mitochondrial disease affecting the kidney Rare Disease Group: This group is to promote the recognition of patients with mitochondrial disease affecting the kidney.
- Monoclonal Gammopathy of Renal Significance Rare Disease Group: To promote the RaDaR registration of patients affected by Monoclonal Gammopathy of Renal Significance (MGRS) To develop standard operating procedures in regards to the treatment of Paraprotein Associated Kidney Diseases To provide better patient information and support To support research, in collaboration with international groups, into basic science, disease progression models and clinical trials
- MPGN, DDD & C3 Glomerulopathy Rare Disease Group: To bring together clinicians, scientists and consumers for the purposes of:
  Undertaking clinical research into the causes of and treatment for MPGN and C3 glomerulopathies Promoting best clinical practice for patients with MPGN and C3 glomerulopathies Facilitating support for patients and families affected by MPGN and C3 glomerulopathies
- Nephrotic Syndrome Rare Disease Group: To compile a comprehensive UK registry of childhood and adult Nephrotic Syndrome, which includes detailed clinical information, laboratory results and genetic testing information where available. The information will be available to the patients/parents, their clinicians, and, in an anonymised form, to the Nephrotic Syndrome Rare Disease Group for research purposes.
  To investigate the underlying cause of Nephrotic Syndrome by comprehensive genetic testing of all patients (with full informed consent), and the study of patient plasma for biomarkers of disease To inform patients about the latest research and educational advances regarding the disease To put patients in touch with recognised support groups and charities To develop treatment and investigation guidelines for clinicians and patients To enable clinical trials to be designed and carried out to further management of the disease
- Pregnancy and Chronic Kidney Disease Rare Disease Group: Increasing numbers of women with chronic kidney disease (CKD) are thinking about pregnancy. It has been known for over 50 years that CKD can affect how a pregnancy progresses and that a pregnancy can have a negative effect on damaged kidneys. However, outcomes have been improving decade by decade.
  The group will develop care pathways for women with CKD throughout pregnancy.
  Specific areas of research interest include:
  What is the best blood pressure target during pregnancy for women with CKD? Is preconception counselling for women with CKD useful? How should we prevent blood clots during pregnancy in women with CKD? What is the effect of protein loss in the urine on pregnancies? Which women with CKD are most likely to develop pre-eclampsia? What is the best way to measure kidney function in pregnant women with CKD? What happens to mothers with CKD and their babies after pregnancy?
- Pure Red Cell Aplasia Rare Disease Group: To increase awareness of Pure Red Cell Aplasia (PRCA). To streamline the diagnostic process. To investigate and implement measures to reduce the incidence of the disease. To empower affected patients in seeking help and support. To establish international collaborations to promote research into the causes and management of the disease.
- Retroperitoneal Fibrosis Rare Disease Group: The Retroperitoneal Fibrosis (RPF) Rare Disease Group aims to:
  establish a registry of patient data and biological samples (plasma, urine, biopsy tissue) collate available information on RPF and develop new information for both patients and carers improve upon observational data in terms of the presentation, natural history and outcomes in RPF patients nationally develop multi-disciplinary consensus care pathways and clinical guidelines for RPF develop a strategy for patient recruitment to trials
- Tuberous Sclerosis Rare Disease Group: There are a number of unanswered questions relating to Tuberous Sclerosis Complex (TSC), which the RDG hopes to be able to address:
  What is the frequency and severity of renal involvement in patients with TSC, particularly as they grow older? What is the frequency of multiple renal AMLs in individuals without other features of TSC? What is the frequency of renal impairment or renal haemorrhage in patients with renal AMLs, and how does this relate the lesion size, number and distribution? What is the frequency of bleeding or renal impairment in patients with multiple renal AMLS treated with mTOR inhibitors or other interventions? What is the frequency of impaired GFR (CKD stage 2 or higher), and what are the causes? What is the efficacy of treatment of renal AMLs in preventing bleeding and preserving GFR? What are the optional treatment regimes with mTOR inhibitors?
- Tubulopathy Rare Disease Group: The newly renamed Tubulopathy Rare Disease Group, previously known as Hypokalaemic Alkaloses, has recently expanded it's inclusion criteria for RaDaR to include a large number of conditions.
- Vasculitis Rare Disease Group: The Vasculitis Rare Disease Group has developed from the UK and Ireland Vasculitis registry initiative UKIVAS. The group members represent Vasculitis units across the UK and participate in Vasculitis research and care.
  We have a number of aims:
  To promote collaboration and sharing of expertise and resources in clinical research
  To develop guidelines for the management of Vasculitis
  To develop a nationwide registry of anonymized demographic, treatment and outcome data for patients with Vasculitis in the UK and Ireland
  To develop high quality patient and clinician information via the Rare Renal and Vasculitis UK websites
  To link with interested patient groups, research collaborations and industry.

SUMMARY:
The goal of this National Registry is to is to collect information from patients with rare kidney diseases, so that it that can be used for research.

The purpose of this research is to:

* Develop Clinical Guidelines for specific rare kidney diseases. These are written recommendations on how to diagnose and treat a medical condition.
* Audit treatments and outcomes. An audit makes checks to see if what should be done is being done and asks if it could be done better.
* Further the development of future treatments.

Participants will be invited to participate on clinical trials and other studies. The registry has the capacity to feedback relevant information to patients and in conjunction with Patient Knows Best (Home - Patients Know Best), allows patients to provide information themselves, including their own reported quality of life and outcome measures.

DETAILED DESCRIPTION:
Background

Rare diseases are arbitrarily defined as having an incidence such that they cannot be studied effectively on patient groups drawn from one or a few medical centres.

A high proportion of such disorders have a genetic background and often these diseases are first expressed in childhood. The success of chronic and end-stage renal failure programmes in childhood permit increased numbers of these patients to survive into adulthood. There are 13 centres for paediatric nephrology in the UK. For a rare disorder that a paediatric nephrologist might diagnosis only once a year, and assuming 100% survival to adulthood, a renal physician might be asked to take over such a case only once in seven or eight years of practice. Research is hampered by this dilution of clinical experience. Similarly in adult practice there are rare complications of diseases or their treatment so that a nephrologist might encounter such an event less often than once in every 5 years. National aggregation of clinical experience is essential to further study.

Research groups investigating a rare disease (Rare Disease Groups, RDGs) have difficulty accessing patients who are widely distributed. While rare disease groups are often successful in identifying novel genotypes in a few individuals, it is more difficult to define phenotype and undertake phenotype-genotype correlations. Moreover, the scarcity of patients makes it difficult to develop biomarkers or identify well-defined cohorts in which to test novel treatments. As a result, the progression and outcome for many rare diseases are unknown and treatment remains underdeveloped.

Purpose

The purpose of the National Registry of Rare Kidney Diseases (RaDaR; rare disease registry) is to facilitate translational and epidemiological research into rare kidney diseases by setting up and maintaining a comprehensive clinical database in partnership with Rare Disease Groups.

RaDaR facilitates the identification of well-characterized cohorts of patients who may be invited to participate in clinical trials, the development of biomarkers, phenotype-genotype correlations or outcome studies. This will inform the development of clinical guidelines for specific rare diseases, audit treatment and outcome and further the development of future therapies.

RaDaR provides an infrastructure to capture both generic and disease-specific clinical information and to collate longitudinal information. Patients and clinicians can view information about the conditions covered by RaDaR on RareRenal.org, which links closely with RaDaR.

RaDaR is predominately aimed at UK patients; however international recruits who are consented in the UK by an NHS hospital are also eligible, subject to local approval.

ELIGIBILITY:
* Kidney Rare Disease
* Paeds and adults
* Eligibility differs for each rare disease group
* See: https://ukkidney.org/rare-renal/recruitment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varies for each Rare Disease Group
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2009-11-06 (Actual); Primary Completion 2039-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Facilitate translational and epidemiological research | 2009-2039
  Setting up and maintaining a comprehensive clinical database in partnership with Rare Disease Groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zoe Plummer, Bristol, South West, United Kingdom